CLINICAL TRIAL: NCT00765245
Title: A Phase II Randomized Study of Lenalidomide or Lenalidomide and Rituximab as Maintenance Therapy Following Standard Chemotherapy for Patients With High/High-intermediate Risk Diffuse Large B-Cell Lymphoma
Brief Title: Lenalidomide With or Without Rituximab After Standard Chemotherapy in Treating Patients With Diffuse Large B-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nishitha Reddy, MD, Assistant Professor of Medicine; Hematologist/Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC HEM 0835; P30CA068485 (NIH)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Lenalidomide (Experimental)
  Interventions: Drug: Lenalidomide
- Arm II: Lenalidomide and Rituximab IV (Experimental): Patients receive lenalidomide as in arm I and rituximab IV on day 8 of courses 1, 3, 5, 7, 9, and 11 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Orally once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Revlimid
  Arms: Arm I: Lenalidomide
Drug: Lenalidomide — Lenalidomide 20 mg daily, Days 1-21, followed by 7 days rest (28-day cycle). Cycles will be repeated every 28 days for a total of 12 cycles
  Other Names: Revlimid
  Arms: Arm II: Lenalidomide and Rituximab IV
Drug: Rituximab — Rituximab 375 mg/m2 intravenously (IV) starting on Day 8, Cycle 1 of lenalidomide. Rituximab will be repeated on Day 8 of odd numbered cycles (Cycles 1, 3, 5, 7, 9, and 11) for a total of 6 doses from randomization.
  Other Names: Rituxan
  Arms: Arm II: Lenalidomide and Rituximab IV

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. It may also stimulate the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether lenalidomide is more effective with or without rituximab in treating diffuse large B-cell non-Hodgkin lymphoma.

PURPOSE: This randomized phase II trial is studying lenalidomide to see how well it works when given with or without rituximab after standard chemotherapy in treating patients with diffuse large B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the 1-year disease-free and relapse-free survival of patients with high- or high/intermediate-risk diffuse large B-cell non-Hodgkin lymphoma treated with maintenance therapy comprising lenalidomide with or without rituximab following standard chemotherapy.

Secondary

* To assess the 2-year disease-free survival of patients treated with these regimens.
* To define the safety and toxicity profile of these regimens.
* To perform antibody-dependent cellular cytotoxicity assays using peripheral blood mononuclear cell samples from these patients.
* To assess the change in the number of natural killer cells by flow cytometric analysis.
* To evaluate cytokines including, but not limited to, sIL-2R, IL-6, IL-15, IL-12, TNF-α, and IFN-γ in these patients.
* To study the KIR genotype receptor and FCγR polymorphisms.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive lenalidomide as in arm I and rituximab IV on day 8 of courses 1, 3, 5, 7, 9, and 11 in the absence of disease progression or unacceptable toxicity.

Peripheral blood mononuclear cells are collected periodically for correlative studies. Samples are analyzed for change in the number of natural killer cells by flow cytometry; antibody-dependent cellular cytotoxicity by assay; cytokines; KIR genotype receptor; and FCγR polymorphisms.

After completion of study therapy, patients are followed at 30 days and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an Informed Consent form
2. Age > 18 years at time of signing the Informed Consent Form
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Patients with histological confirmation of diffuse large B cell lymphoma with at least one of the following characteristics:

   * High or intermediate IPI score (See Appendix 8.0 for IPI scoring criteria)
   * Patients who are still PET scan positive mid therapy with R-CHOP, but, have turned negative after completion of therapy.
   * Low risk International prognostic index ie., an IPI score of <3 if age >60 years or <2 if age is less than or equal to 60 with c-myc positive by Fluorescent In situ Hybridization.
5. No other previous lymphoma therapy, hormonal therapy or surgery, except for standard therapy with R-CHOP with or without radiation and with or without prophylactic Methotrexate therapy. Patients must be enrolled within 4-12 weeks of completion of therapy.
6. At the time of study entry following standard therapy with R-CHOP±RT, patients should be in complete remission.
7. ECOG performance status of ≤ 2 at study entry
8. Laboratory test results within these ranges:

   * Absolute neutrophil count ≥ 1500/mm³
   * Platelet count ≥100K /mm³
   * Serum creatinine ≤ 2.0 mg/dL
   * Total bilirubin ≤ 1.5 mg/dL
   * AST (SGOT) and ALT (SGPT) ≤ 2 x ULN
9. Disease free of prior malignancies for ≥ 3 years with exception of currently treated basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
10. All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the Revlimid REMS® program.

    •Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by the Revlimid REMS® program) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
11. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation, if patients are thought to be at an elevated risk of thrombosis.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the Informed Consent
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. Concurrent use of other anti-cancer agents or treatments.
9. Known positive for HIV or infectious hepatitis, type B or C.
10. A diagnosis of deep vein thromboses in the preceding 3 months of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nishitha Reddy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Vose JM, Habermann TM, Czuczman MS, Zinzani PL, Reeder CB, Tuscano JM, Lossos IS, Li J, Pietronigro D, Witzig TE. Single-agent lenalidomide is active in patients with relapsed or refractory aggressive non-Hodgkin lymphoma who received prior stem cell transplantation. Br J Haematol. 2013 Sep;162(5):639-47. doi: 10.1111/bjh.12449. Epub 2013 Jul 9. PMID 23834234
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study began enrolling patients October 2008 and continued until November 2013 when its study accrual goal was met. Patients were recruited from two academic medical institutions, Vanderbilt University Medical Center, Vanderbilt-Ingram Cancer Center and the University of North Carolina Medical Center, Chapel Hill.
Pre-assignment Details: Fifty-one patients signed consent to participate in this trial. Seven patients did not meet eligibility criteria, thus they did not receive treatment therapy and continue on study.
Period: Overall Study
Arm/Group | Arm I: Lenalidomide | Arm II: Lenalidomide and Rituximab IV
Started | 22 | 22
Completed | 9 | 20
Not Completed | 13 | 2
Not completed — disease progression | 3 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Lenalidomide | Arm II: Lenalidomide and Rituximab IV | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 32
  >=65 years | 7 | 5 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [54.8 to 69.5] | 59.0 [49.5 to 62.5] | 59 [52 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 18 | 38
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 19 | 18 | 37
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival at 1 Year
Description: Disease-free survival is the time from on-treatment to first relapse or death (whichever comes first). Those who are alive and without relapse are censored at the last date known alive.
Time Frame: From on-treatment date to disease recurrence, up to 1 year
Measure: Mean (95% Confidence Interval); unit: years
Arm/Group | Arm I: Lenalidomide | Arm II: Lenalidomide and Rituximab IV
Number analyzed (Participants) | 22 | 22
years | 0.818 [0.58 to 0.94] | 0.90 [0.58 to 0.94]

2. Secondary Outcome: Disease-free Survival at 2 Years
Description: Disease-free survival is the estimated probable duration of life from on-study date to date of death from any cause, using the Kaplan-Meier method where death is an event, with censoring for non-expired patients at last known date alive.
Time Frame: From on-treatment date to disease recurrence, up to 2 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I: Lenalidomide | Arm II: Lenalidomide and Rituximab IV
Number analyzed (Participants) | 22 | 22
years | 0.818 [0.585 to 0.928] | 0.757 [0.506 to 0.893]

3. Secondary Outcome: Number of Patients With Each Worst-Grade Toxicity
Description: Count of patients according to the worst-grade toxicity experienced by each, where worst-grade toxicity is per NCI common toxicity criteria: grade 1, mild; grade 2, moderate; grade 3, severe; grade 4, life-threatening; grade 5, death. Toxicities present at baseline and continuing without change in grade are excluded when considering worst-grade toxicity.
Time Frame: 30 days after completing treatment, for up to 13 months
Population: Total number of patients reported with any toxicity
Measure: Number; unit: participants
Arm/Group | Arm I: Lenalidomide | Arm II: Lenalidomide and Rituximab IV
Number analyzed (Participants) | 19 | 21
participants
  Number of patients with WGT=1 | 2 | 0
  Number of patients with WGT=2 | 6 | 8
  Number of patients with WGT=3 | 6 | 8
  Number of patients with WGT=4 | 5 | 5
  Number of patients with WGT=5 | 0 | 0

4. Other Pre Specified Outcome: Investigate Potential Predictive Biomarkers of Clinical Response or Resistance to Lenalidomide
Time Frame: up to two years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Exploratory: Concordance Between IHC for GCB and Non-GCB Subtypes to the Gene Expression Profiles Associated With the Subtypes
Time Frame: up to two years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days after completing treatment (up to 13 months).
Arm/Group | Arm I: Lenalidomide | Arm II: Lenalidomide and Rituximab IV
Serious Adverse Events (participants affected / at risk) | 8/22 | 1/22
Other Adverse Events (participants affected / at risk) | 22/22 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Lenalidomide (N=22) | Arm II: Lenalidomide and Rituximab IV (N=22)
Pain - headache (Nervous system disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Speech impairment (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0)
Obstruction - ureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (Investigations) | 2 (2) | 0 (0)
Fever (in the absence of neutropenia) (General disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection (Investigations) | 1 (2) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0)
Secondary Malignancy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction - small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Lenalidomide (N=22) | Arm II: Lenalidomide and Rituximab IV (N=22)
hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (10)
ALT, SGPT (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
AST, SGOT (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
ataxia - incooridnation (Nervous system disorders) | 1 (1) | 0 (0)
auditory - other (Ear and labyrinth disorders) | 1 (1) | 0 (0)
bruising (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
hypercholesteremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
confusion (Psychiatric disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 7 (10) | 7 (8)
cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (12)
creatinine (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
dehydration (Gastrointestinal disorders) | 1 (1) | 1 (1)
peridontal disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
dermatology - other (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (5)
diarrhea (Gastrointestinal disorders) | 9 (11) | 11 (13)
Distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 1 (1)
xerostomia (dry mouth) (Gastrointestinal disorders) | 3 (3) | 5 (5)
dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (8)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
edema (General disorders) | 5 (7) | 5 (8)
gait/walking disturbance (Gastrointestinal disorders) | 2 (2) | 0 (0)
fatigue (General disorders) | 14 (15) | 13 (15)
fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
gastrointestinal - other (Gastrointestinal disorders) | 5 (6) | 5 (5)
hyperglycemia (Metabolism and nutrition disorders) | 4 (6) | 2 (2)
dyspepsia (heartburn) (Gastrointestinal disorders) | 3 (3) | 2 (2)
hemoglobin increase (Investigations) | 5 (5) | 5 (5)
hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
hypertension (Vascular disorders) | 2 (2) | 2 (2)
incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
infection (Infections and infestations) | 13 (14) | 15 (18)
Insomnia (Psychiatric disorders) | 6 (6) | 6 (6)
joint function (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
laryngeal nerve dysfunction (Nervous system disorders) | 1 (1) | 1 (1)
leukocytes (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
memory impairment (Nervous system disorders) | 0 (0) | 2 (2)
metabolic other (Metabolism and nutrition disorders) | 2 (3) | 3 (4)
mood alteration (Psychiatric disorders) | 6 (7) | 1 (2)
musculoskeletal soft tissue (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1) | 5 (7)
neuropathy (Nervous system disorders) | 8 (10) | 11 (16)
neutrophil count increased (Investigations) | 9 (13) | 11 (15)
pain - abdomen (General disorders) | 7 (8) | 0 (0)
pain - back (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
pain - chest wall (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
pain - extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
pain - headache (Nervous system disorders) | 4 (5) | 8 (9)
pain - joint (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
pain - other, NOS (General disorders) | 2 (2) | 4 (4)
hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
desquamation - rash (Skin and subcutaneous tissue disorders) | 11 (13) | 6 (9)
acne/acneiform (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (5)
renal - other (Renal and urinary disorders) | 1 (1) | 1 (1)
rigors (General disorders) | 1 (1) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
dysgeusia (Gastrointestinal disorders) | 2 (2) | 0 (0)
hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2)
hypothyroidism (Endocrine disorders) | 2 (2) | 4 (4)
urinary frequency (Renal and urinary disorders) | 1 (1) | 3 (3)
urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
blurred vision (Eye disorders) | 1 (1) | 1 (1)
dysarthria (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
vomiting (Gastrointestinal disorders) | 7 (8) | 5 (6)
non-infectious wound complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
"Pre-specified Outcomes Measures" data were not collected as anticipated in original protocol, thus results will not be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes